CLINICAL TRIAL: NCT05736978
Title: Clinical Efficacy and Safety of Adaptive Treatment of Acute Myeloid Leukemia (AML) Based on D14 MRD results-a Multicenter, Single-arm, Prospective Clinical Study
Brief Title: Adaptive Treatment for Acute Myeloid Leukemia Based on D14 MRD Results
Acronym: AVS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Tong Ren Hospital (Other)
Responsible Party: Principal Investigator, Liu Ligen, director, Shanghai Tong Ren Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AVS
Record Dates: First submitted 2023-02-12; First posted 2023-02-21 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: AML; MRD
Keywords: untreated AML; MRD results; selinexor
MeSH Terms: interventions — Azacitidine; venetoclax; selinexor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment regimen based on C1D14 MRD (Experimental): Untreated acute myeloid leukemia who are ineligible for intensive chemotherapy will be given azacitidine 75mg/m2, d1-7 and venetoclax 100mg on day 1 and 200mg on day 2, 400mg on day 3-28. Based on MRD results on C1D14, MRD negative patients will go on azacitidine and venetoclax regimen and for patients with MRD positive, selinexor 60mg on D15 and D22 will be added. Patients can receive transplants at any time once they achieved complete remission and other patients will continue to receive treatment until disease progression or unacceptable toxic effects.
  Interventions: Drug: Azacitidine; Drug: Venetoclax; Drug: Selinexor

INTERVENTIONS:
Drug: Azacitidine — 75mg/m2 d1-7
Drug: Venetoclax — d1 100mg, d2 200mg, d3-28 400mg
  Other Names: ABT-199
Drug: Selinexor — if MRD positive in C1D14, selinexor 60mg D15, D22
  Other Names: XPO1 inhibitor

SUMMARY:
This is a prospective, single-arm, multi-center clinical trial to evaluate the efficacy and safety of selinexor in combination with azacitidine and venetoclax for untreated acute myeloid leukemia based on MRD results on day 14 of the first cycle.

DETAILED DESCRIPTION:
Azacitidine and Venetoclax will be given at the approved dose regimen for 75mg/m2, d1-7(azacitidine) and 100mg on day 1 and 200mg on day 2, 400mg on day 3-28 (venetoclax), 28 days per cycle. Based on MRD results on C1D14, MRD negative patients will go on azacitidine and venetoclax regimen and for patients with MRD positive, selinexor 60mg on D15 and D22 will be added. Patients can receive transplants at any time once they achieved complete remission and other patients will continue to receive treatment until disease progression or unacceptable toxic effects.

ELIGIBILITY:
Inclusion Criteria:

* Known and written informed consent voluntarily
* Age ≥ 18 years
* Newly diagnosed AML patients (per WHO 2022 classification criteria for AML diagnosis), who are not suitable for intensive chemotherapy:

  * 75 years or Aged 18 to 74 years with at least one of the following comorbidities: Eastern Cooperative Oncology Group (ECOG) performance status score of 2 or 3 or 4; Cardiac history of Congestive Heart Failure (CHF) requiring treatment or Ejection Fraction <= 50% or chronic stable angina; Diffusing capacity of the Lung for Carbon Monoxide (DLCO) <= 65% or Forced Expiratory Volume in 1 second (FEV1) <= 65%; Creatinine clearance >= 30 mL/min to < 45 ml/min; Moderate hepatic impairment with total bilirubin > 1.5 to <= 3.0 × Upper Limit of Normal (ULN); Any other comorbidity that the physician judges to be incompatible with intensive chemotherapy .
* Liver function meets the following criteria: aspartate aminotransferase (AST) ≤ 3.0×ULN*; alanine aminotransferase (ALT) ≤3.0×ULN*; Bilirubin≤1.5×ULN*; For subjects <75 years old, the bilirubin level can be ≤3.0×ULN; Unless due to leukemic organ involvement.
* Renal function meets the following criteria: creatinine clearance ≥ 30 mL/min (Cockroft-Gault formula)
* Life expectancy ≥ 4 weeks

Exclusion Criteria:

* History of any malignancies prior to study entry with exception noted in the protocol.
* Participant has known HIV infection, active hepatitis B virus (HBV) and/or hepatitis C virus (HCV) .
* Participant has known active central nervous system (CNS) involvement with AML.
* Must not have received prior anti-AML treatment except for hydroxyurea

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2023-03-31 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2027-03-15 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With Composite Complete Remission | From the study start up to death (up to approximately 2 years; )

SECONDARY OUTCOMES:
overall survival (OS) | From the study start up to death (up to approximately 4 years; )
Overall response rate(ORR) | From the study start up to death (up to approximately 4 years; )
percentage of patients who achieved MRD negativity | From the study start up to death (up to approximately 4 years; )
Recurrence Free Survival(RFS) | From the study start up to death (up to approximately 4 years; )

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Beizhan Hospital, Shanghai
  - Pla Navy Feature Medical Center, Shanghai
  - Shanghai Ruijin Hospital, Shanghai
  - Shanghai Tong Ren hospital, Shanghai

IPD SHARING:
Plan to Share IPD: No